CLINICAL TRIAL: NCT01878929
Title: The Effect of Pollen Season on Subcutaneous Allergen Immunotherapy Reactions: A Double Blind Randomized Control Trial.
Brief Title: The Effect of Pollen Season on Subcutaneous Allergen Immunotherapy Reactions
Acronym: SCIT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Devi Jhaveri, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-13-06
Record Dates: First submitted 2013-05-28; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Allergic Rhinitis; Asthma; Allergic Conjunctivitis
Keywords: pollen; allergen immunotherapy; subcutaneous allergen immunotherapy; SCIT
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Conjunctivitis, Allergic | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allergen(Tree, Grass, Weeds) -Held (Active Comparator): Allergen(Tree, Grass, Weeds)-Held
  Weekly administration of Greer manufactured allergen extract at same dose and concentration patient was on prior to allergen season for the duration of patients allergen season.
  Interventions: Drug: Allergen(Tree, Grass, Weeds)
- Allergen(Tree, Grass, Weeds) -Build-up (Active Comparator): Allergen(Tree, Grass, Weeds) -Build-up
  Weekly administration of Greer manufactured allergen extract at escalating dose and concentration patient for the duration of patients allergen season.
  Interventions: Drug: Allergen(Tree, Grass, Weeds)

INTERVENTIONS:
Drug: Allergen(Tree, Grass, Weeds) — Greer is manufacture of all allergen extract used in this study.
  Other Names: "Greer Grass Extract"; "Greer Tree Extract"; "Greer Ragweed Extract"; "Greer Weed Extract"; "Greer Tree and Ragweed Extract"; "Greer Grass and Ragweed Extract"; "Greer Weed and Ragweed Extract"; "Greer Tree and Grass Extract"; "Greer Weed and Grass Extract"; "Greer Weed and Tree Extract"; "Greer Tree and Grass and Ragweed Extract"; "Greer Grass and Ragweed and Weed Extract"; "Greer Tree and Ragweed and Weed Extract"; "Greer Tree and Grass and Weed Extract"; "Greer Tree and Grass and Ragweed and Weed Extract"

SUMMARY:
Subcutaneous allergen immunotherapy (SCIT) is a widely used and effective treatment modality for allergic rhinoconjunctivitis and asthma. SCIT starts with a build-up phase during which a patient receives frequent, escalating doses of the allergens they are allergic to until they reach a predetermined maintenance dose. This is followed by a maintenance phase during which the allergen dose is kept constant and administered at greater intervals. Maximum clinical improvement is generally not seen until a patient is in the maintenance phase. Anecdotal evidence of possible reactions to SCIT administered during a patient's pollen season has led to dosage freezes during a patient's pollen season which extends the length of the build-up phase by many months. Prolonging the buildup phase increases the time required to obtain maximal benefit from SCIT, and at the same time, can decrease patient compliance with therapy due to the prolonged period of time when frequent injections are required.

The aims of this study are to determine if adverse reactions to pollen SCIT are increased if doses are increased during pollen season.

DETAILED DESCRIPTION:
Subcutaneous allergen immunotherapy (SCIT) is a widely used and effective treatment modality for allergic rhinoconjunctivitis and asthma. SCIT starts with a build-up phase during which a patient receives frequent, escalating doses of the allergens they are allergic to until they reach a predetermined maintenance dose. This is followed by a maintenance phase during which the allergen dose is kept constant and administered at greater intervals. Maximum clinical improvement is generally not seen until a patient is in the maintenance phase. Anecdotal evidence of possible reactions to SCIT administered during a patient's pollen season has led to dosage freezes during a patient's pollen season which extends the length of the build-up phase by many months. Prolonging the buildup phase increases the time required to obtain maximal benefit from SCIT, and at the same time, can decrease patient compliance with therapy due to the prolonged period of time when frequent injections are required.

The aims of this study are to determine if adverse reactions to pollen SCIT are increased if doses are increased during pollen season.

Specific Aim 1: To determine if escalating pollen SCIT doses during the pollen season is associated with an increased rate of immediate reactions in comparison to holding SCIT doses constant.

Hypothesis: There will not be an increased rate of immediate reactions to SCIT in build up phase received during the pollen season in comparison to SCIT held for pollen season.

Strategy: In a prospective trial, 245 subjects will be randomized to receive monthly (doses held constant) or weekly (doses built up) injections. Rate of immediate local and systemic reactions per injection will be compared between the two groups.

Specific Aim 2: To determine if escalating pollen SCIT doses during the pollen season is associated with an increased rate of delayed reactions in comparison to holding SCIT doses constant.

Hypothesis: There will not be an increased rate of delayed reactions to SCIT in build up phase received during the pollen season in comparison to SCIT held for pollen season.

Strategy: In a prospective trial, 245 subjects will be randomized to receive monthly (doses held constant) or weekly (doses built up) injections. Rate of delayed reactions per injection will be compared between the two groups.

BACKGROUND AND SIGNIFICANCE

Immunotherapy is one of the most effective therapies for allergic rhinoconjunctivitis, but the protocol dosing during pollen season is based on limited data. Immunotherapy is given in increasing dosage during the build up phase in order to build tolerance. After the build up phase, there is a maintenance phase that is used for the remainder of therapy. At this time, there is little data to support the common practice of not increasing the dosage of immunotherapy during pollen seasons.

The recent allergen immunotherapy practice parameter references 2 articles that have noted no increased systemic reactions to SCIT during pollen season. , In one prospective study, it was concluded that there was no direct correlation of reactions to SCIT and pollen season.3 They did note a correlation between the mean monthly mold counts in August to October and the rate of systemic reactions. The other study referenced is a prospective study which did not observe a statistically significant difference in the rate of systemic reactions to grass or ragweed pollen during their respective pollen seasons.4 However, the conclusions of these studies are conflicted by another study which consists of surveys retrospectively sent to members of the American Academy of Allergy Asthma and Immunology. The surveys in this study identified 46% of near fatal reactions to SCIT as occurring during peak allergy season. Though the immunotherapy standard parameters are not defining pollen season as a contraindication, we will consider it more that minimal risk for this study.

It is still common practice to stop the buildup phase and not escalate SCIT dosing during pollen season due to the conflicting available data and limitations in study design of many of the studies (retrospective, questionnaire based). A further look into SCIT dosing during pollen season will allow for more standardized practice and potentially improved patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* include individuals ages 5 and greater at Allergy/Immunology Associates, Inc., who are receiving build-up SCIT to tree, grass, and/or weed pollens for allergic rhinitis, allergic conjunctivitis, and/or asthma

Exclusion Criteria:

1. are in maintenance phase of SCIT
2. are on beta-blockers
3. have a forced expiratory volume in 1 second (FEV1) of less than 70% of predicted
4. have a history of anaphylaxis with previous SCIT to aeroallergens (as defined by the requirement of intramuscular or subcutaneous epinephrine for treatment of a SCIT-induced reaction)
5. have any uncontrolled cardiac or pulmonary disease as determined by their treating allergist/immunologist
6. are pregnant, due to risk of harm to fetus if anaphylaxis occurs.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Immediate Reaction Rate of Build-Up Phase in Pollen Season | 1 year
  To determine if escalating pollen SCIT doses during the pollen season is associated with an increased rate of immediate reactions in comparison to holding SCIT doses constant.

SECONDARY OUTCOMES:
Delayed Reaction Rate of Build-Up Phase during Pollen Season | 1 year.
  To determine if escalating pollen SCIT doses during the pollen season is associated with an increased rate of delayed reactions in comparison to holding SCIT doses constant.

CONTACTS AND LOCATIONS:
Overall Officials: Devi K Jhaveri, D.O., Principal Investigator — University Hospitals Cleveland Medical Center; Haig Tcheurekdjian, M.D., Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Allergy/Immunology Associates Inc., South Euclid, Ohio, United States